CLINICAL TRIAL: NCT01163006
Title: Soluble Dietary Fibres as Dietetic Aid to Reduce the Risks of Type 2 Diabetes Mellitus
Brief Title: Soluble Dietary Fibres in the Prevention of Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Tate and Lyle Ingredients France (Industry)
Responsible Party: Sponsor
Other Study IDs: MEC 09-3-084
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2010-07

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — polydextrose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- polydextrose (Experimental)
  Interventions: Other: Polydextrose and soluble gluco fibre
- soluble glucofibre (Experimental)
  Interventions: Other: Polydextrose and soluble gluco fibre
- isocaloric dietary control (Placebo Comparator)
  Interventions: Other: Polydextrose and soluble gluco fibre
- full caloric control (Placebo Comparator)
  Interventions: Other: Polydextrose and soluble gluco fibre

INTERVENTIONS:
Other: Polydextrose and soluble gluco fibre — Polydextrose and soluble gluco fibre

SUMMARY:
Controlling the glycemic impact of foodstuffs (by reducing the glycemic load of the diet by using soluble dietary fibres) may reduce the glycemic or insulinemic response. This may in turn result in a reduced inhibition of postprandial fat oxidation rate and a lower plasma triacylglycerol concentration A higher postprandial fat oxidation may result in less lipid accumulation in non-adipose tissue thereby improving insulin sensitivity and the metabolic profile in the longer term.

ELIGIBILITY:
Inclusion Criteria:

* Overweight men and women

Exclusion Criteria:

* regular smokers, athletes, diabetes mellitus

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
fat oxidation

SECONDARY OUTCOMES:
24h glucose pattern

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Netherlands